CLINICAL TRIAL: NCT05641168
Title: A Pilot Evaluation Exploring New Adhesive Materials and Their Ability to Adhere to Abdominal and Peristomal Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CP333
Record Dates: First submitted 2022-11-15; First posted 2022-12-07 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Skin Abnormalities
MeSH Terms: conditions — Skin Abnormalities | interventions — Adhesives

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ostomy Adhesive material (Experimental): Newly designed ostomy adhesive material
  Interventions: Other: Adhesive material
- comparator adhesive material (Other): Adhesive material already on the market e.g adhesive material from SenSura Mio ostomy product
  Interventions: Other: Standard adhesive material

INTERVENTIONS:
Other: Adhesive material — Newly developed adhesive material
  Arms: Ostomy Adhesive material
Other: Standard adhesive material — Standard adhesive material
  Arms: comparator adhesive material

SUMMARY:
The study investigates different adhesive materials on healthy and peristomal skin

ELIGIBILITY:
Inclusion Criteria:

* Has given written consent
* Be at least 18 years of age and have full legal capacity
* Have had a colostomy/ileostomy/urostomy for more than one year (for stoma patients) Have suitable peristomal skin area (assessed by investigator) (for stoma patients)

Exclusion Criteria:

* Currently receiving or have within the past 2 months received radio- and/or chemotherapy
* Currently receiving or have within the past month received topical steroid treatment in the abdominal skin area or systemic steroid (tablet/injection) treatment
* Are pregnant or breastfeeding
* Having dermatological problems in the abdominal area (assessed by investigator)
* Participate in other clinical investigations. Exception: Participation in other Coloplast sponsored clinical investigations is accepted under the circumstances that the subject has paused the activities in the investigation and are otherwise complying with the inclusion and exclusion criteria of this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Adherent area | At every material change throughout the study, an average of 1 week
  Adherent area (assessed by photos of adhesive materials)

CONTACTS AND LOCATIONS:
Locations (1):
- Coloplast Research Unit/Userlab, Humlebæk, Denmark